CLINICAL TRIAL: NCT02368327
Title: Clinical Study to Generate Exploratory Training Set of Data on the Time Course of Gene Expression Profile at Site of Antigen Deposition Compared With Whole Blood Following IM Injection With Alum or MF59-adjuvanted Protein Subunit Vaccines
Brief Title: Gene Expression Profiles in Muscle After Immunisation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Surrey (Other)
Collaborators: Max Planck Institute for Infection Biology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: CRC305E
Record Dates: First submitted 2015-02-13; First posted 2015-02-23 (Estimated); Last update posted 2015-08-10 (Estimated); Status verified 2015-02

CONDITIONS: Healthy
MeSH Terms: interventions — fluad vaccine; Fendrix

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (3):
- Fluad (Active Comparator): Participants receive one dose of Fluad vaccine
  Interventions: Biological: Fluad
- Fendrix (Active Comparator): Participants receive one dose of Fendrix vaccine
  Interventions: Biological: Fendrix
- Placebo (Placebo Comparator): Participants receive one dose of saline placebo
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Fluad
  Arms: Fluad
Biological: Fendrix
  Arms: Fendrix
Biological: Placebo
  Arms: Placebo

SUMMARY:
This clinical study is part of the BIOVACSAFE project which is funded by the Innovative Medicine Initiative. In this study we will take a small muscle biopsy in order to identify any differences in the response around the actual site of injection compared with responses we measure in blood at the same time.

ELIGIBILITY:
Inclusion Criteria:

1. The participant is able to read and understand the Informed Consent Form (ICF), and understand study procedures.
2. The participant has signed the ICF.
3. Healthy male participants aged 18-45 years inclusive.
4. BMI between 19-27 kg/m2.
5. Pre-immunised with Hepatitis B vaccine
6. Hepatitis B sAb positive (evidence of vaccine-induced immunity)
7. Hepatitis B sAg and cAb negative (evidence of lack of prior/current HBV infection)
8. Hepatitis C and HIV seronegative.
9. Available for follow-up for the duration of the study.
10. Agree to abstain from donating blood during the study.
11. The participant is, in the opinion of the investigator, healthy on the basis of a, medical history, a symptom directed medical examination and vital signs.

Exclusion Criteria:

1. History of hypersensitivity to any of the vaccine components or a history of any allergy that in the opinion of the investigator would contraindicate participant participation
2. Clinically significant psychiatric, cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, neurological (particularly myasthenia gravis), immunological, or haematological disease or abnormality, as determined by the study physician.
3. Known immune or coagulation disorder or clinically significant abnormalities of platelets, Hb or coagulation on screening labs
4. Known allergy to injected local anaesthetics
5. Unwilling to undergo muscle biopsies
6. Use of steroids or immunosuppressive/immunomodulating drugs either orally or parenterally within 3 months of visit 1.
7. Currently participating in a clinical trial with an investigational or non- investigational drug or device, or has participated in another clinical trial within the 3 months preceding the study.
8. Any condition that, in the investigator's opinion, compromises the participant's ability to meet protocol requirements or to complete the study.
9. Receipt of blood products or immunoglobin, within 3 months of visit 1.
10. Unable to read and speak English to a fluency level adequate for the full comprehension of procedures required in participation and consent.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2015-02; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline values of gene expression in whole blood and muscle | Day 0, Day 0+3 hours, Day 1, Day 3, Day 5 and Day 7

CONTACTS AND LOCATIONS:
Overall Officials: Aldona Greenwood, Principal Investigator — University of Surrey
Locations (1):
- Surrey Clinical Research Centre, Guildford, Surrey, United Kingdom